CLINICAL TRIAL: NCT03287973
Title: Effect of Weight Loss and CPAP on OSA and Metabolic Profile Stratified by Craniofacial Phenotype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Susanna SS Ng, Honorary assistant professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OSA-Craniofacial study
Record Dates: First submitted 2017-09-14; First posted 2017-09-19 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research assistant who scores the sleep study and the laboratory technician who does the blood test are blinded to the intervention arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle modification program group (Active Comparator): Patients with apnea-hypopnea index (AHI) ≥ 15/hr on home sleep study will participate in a dietitian-led lifestyle modification program (LMP) for 6 months. Patients will attend dietary consultation weekly in the first 4 months, and then monthly in the following two months.
  Interventions: Behavioral: Lifestyle modification
- CPAP group (Other): Patients randomized into the continuous positive airway pressure (CPAP) group in each arm will be interviewed by the physician on duty and invited to start autoCPAP treatment for 6 months. They will be offered a CPAP education package. Patients will then commence autoCPAP treatment for 6 months at home.
  Interventions: Device: Continuous positive airway pressure (CPAP)

INTERVENTIONS:
Behavioral: Lifestyle modification — A caloric reduction of 10-20% in daily energy intake from the patient's usual diet (i.e. a deficit ≥ 200 calories per day) will be set as the general initial goal, which will be adjusted subsequently based on changes in body weight with target body mass index (BMI) towards 23 kg/m2.
  Arms: Lifestyle modification program group
Device: Continuous positive airway pressure (CPAP) — Patients randomized into the continuous positive airway pressure (CPAP) group in each arm will be interviewed by the physician on duty and invited to start autoCPAP treatment for 6 months. They will be offered a CPAP education package. Patients will then commence autoCPAP treatment for 6 months at home.
  Arms: CPAP group

SUMMARY:
Obstructive sleep apnea (OSA) is a common form of sleep-disordered breathing (SDB). Weight reduction has always been advocated in patients with OSA who are overweight and may lead to improvement in the severity of OSA. Previous study reported a randomized controlled trial of dietician-led lifestyle modification program (LMP) in 104 patients and found that LMP group had significantly more weight loss and reduced OSA severity, and the response was sustained after 8 months.

This study is aimed to compare the effect of weight loss or CPAP alone on subclinical inflammation, insulin resistance and blood pressure in patients with obesity and moderate-to-severe obstructive sleep apnea, stratified according to the degree of craniofacial restriction.

The study plans to recruit consecutive patients who have been referred to the Respiratory Clinic at the Prince of Wales Hospital with clinical suspicion of sleep-disordered breathing with specific study entry criteria including an age of 18 or more, body mass index (BMI) >25 kg/m2, and moderate to severe OSA diagnosed by home sleep study. Patients having conditions that will affect the serum level of hsCRP will be excluded.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common form of sleep-disordered breathing (SDB). It causes sleep fragmentation, disabling daytime sleepiness, impaired cognitive function, poor quality of life and cardiovascular diseases. Weight reduction has always been advocated in patients with OSA who are overweight and may lead to improvement in the severity of OSA. Previous study reported a randomized controlled trial of dietician-led lifestyle modification program (LMP) in 104 patients and found that LMP group had significantly more weight loss and reduced OSA severity, and the response was sustained after 8 months. However, a wide variety of response to the therapy was observed with 21.3% of patients with severe disease that converted to mild to moderate and only 6.6% of those with severe disease who became mild in severity. Apart from obesity, craniofacial factors are well recognized in the pathogenesis of OSA and are likely to play an important role in influencing the response to weight loss. For the same degree of OSA severity, Caucasians were more overweight whereas Chinese exhibited more craniofacial bony restriction. Recent studies showed that a smaller craniofacial skeleton is associated with better response from weight loss program in terms of OSA improvement. With vast majority of studies investigating the cardiometabolic changes after CPAP or weight loss on patients with OSA, evaluation based on craniofacial restriction, the key factor in the pathogenesis, is lacking.

This study aimed to compare the effect of weight loss or CPAP alone on subclinical inflammation, insulin resistance and blood pressure in patients with obesity and moderate-to-severe obstructive sleep apnea, stratified according to the degree of craniofacial restriction.

The study plans to recruit consecutive patients who have been referred to the Respiratory Clinic at the Prince of Wales Hospital with clinical suspicion of sleep-disordered breathing with specific study entry criteria including an age of 18 or more, body mass index (BMI) >25 kg/m2, and moderate to severe OSA diagnosed by home sleep study. Patients having conditions that will affect the serum level of hsCRP will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with moderate or severe obstructive sleep apnea ( apnea hypopnea index (AHI) ≥ 15); body mass index ≥25 kg/m2; age 18-70 years.

Exclusion Criteria:

* Predominant central sleep apnea; conditions that will affect the level of hsCRP; unstable cardiovascular disease (e.g. recent unstable angina, myocardial infarction, stroke or transient ischemic attack within the previous 6 months or severe left ventricular failure; neuromuscular disease affecting or potentially affecting respiratory muscles; moderate to severe respiratory disease (i.e. breathlessness affecting activities of daily living) or documented hypoxemia or awake SaO2 <92%); psychiatric disease that limits the ability to give informed consent or complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
changes in hsCRP | 6 months

SECONDARY OUTCOMES:
change in Epworth Sleepiness Scale (ESS) | 6 months
Change of insulin sensitivity by Matsuda index | 6 months
Change of facial measurements on photography | 6 months
  Frontal and profile digital photographs of the head and neck are obtained with a standardized setup. A digital camera is mounted on a tripod at a distance of 160 cm from the subject alignment plane.
  Subjects are photographed standing upright while assuming the natural head position. Standardized methods are used to align subjects for the photographs. For the frontal photograph, the subject's facial landmark nasion is aligned along the subject alignment plane while ensuring both ears are seen equally from the front. For the profile photograph, the subject is instructed to turn 90 degrees to the left after the frontal photograph was taken.
  The subject's mid-sagittal plane is aligned to the subject alignment plane. Using image analysis software (Image J v1.36, NIH, Bethesda, MD), the photographs are examined for landmark digitization.
Change of anatomic measurements of upper airway on computed tomography imaging | 6 months
  All subjects will perform a three-dimensional (3D) computed tomography (CT) scans of the head/neck region to evaluate the size of the maxillomandibular volume (MMV) based on the mandibular cephalometric landmarks (left and right condylion, left and right gonion, and menton). All measurements will be made by a single assessor and the analysis will be performed blind to knowledge of AHI data.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna SS Ng, MBChB, Principal Investigator — Chinese University of Hong Kong; Susanna Ng, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ng SSS, Tam WWS, Lee RWW, Chan TO, Yiu K, Yuen BTY, Wong KT, Woo J, Ma RCW, Chan KKP, Ko FWS, Cistulli PA, Hui DS. Effect of Weight Loss and Continuous Positive Airway Pressure on Obstructive Sleep Apnea and Metabolic Profile Stratified by Craniofacial Phenotype: A Randomized Clinical Trial. Am J Respir Crit Care Med. 2022 Mar 15;205(6):711-720. doi: 10.1164/rccm.202106-1401OC. PMID 34936531